CLINICAL TRIAL: NCT07111312
Title: Placebo-controlled, Parallel, Randomized (1:1), Double-blind Study Over 6 Months to Evaluate the Efficacy and Safety of the Food Supplement Olistic Women.
Brief Title: Clinical Evaluation of a Nutraceutical Supplement (Olistic Women) for Hair Growth and Hair Loss in Human Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olistic Research Labs S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-OW-02
Record Dates: First submitted 2025-07-31; First posted 2025-08-08 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Telogen Effluvium
MeSH Terms: interventions — Minerals; Plant Extracts

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Product Arm (Active Comparator)
  Interventions: Dietary Supplement: Drinkable multifactorial food supplement containing vitamins, minerals, plant extracts, and other bioactive compounds, formulated to support hair growth and scalp health in women.
- Placebo Arm (Placebo Comparator)
  Interventions: Other: Placebo control

INTERVENTIONS:
Dietary Supplement: Drinkable multifactorial food supplement containing vitamins, minerals, plant extracts, and other bioactive compounds, formulated to support hair growth and scalp health in women. — Drinkable multifactorial food supplement in liquid form, administered once daily in a 25 mL single-dose vial, for a duration of 180 days. The formulation contains a combination of vitamins, minerals, plant extracts, amino acids, and other bioactive compounds designed to support hair growth and scalp health in women.
  Arms: Active Product Arm
Other: Placebo control — Drinkable formulation consisting of an excipient formulation designed to mimic the organoleptic properties of the active product, reproducing its color and texture while achieving a highly similar taste profile.
  Arms: Placebo Arm

SUMMARY:
Hair loss is a multifactorial and complex condition influenced by factors such as hormonal changes, vitamin and mineral deficiencies, genetic predisposition, oxidative stress, aging, inflammation, and psychological stress. This 6-month randomized, double-blind, placebo-controlled study aimed to evaluate the efficacy and safety of a drinkable nutraceutical formulated with natural, high-quality, patented, and standardized ingredients designed to support hair health through multiple biological pathways. A total of 106 premenopausal women aged 18 to 40 years and diagnosed with telogen effluvium were randomized to receive either the nutraceutical (n = 53) or placebo (n = 53). The primary endpoint was the increase in hair density from baseline versus placebo. The secondary endpoint was the change in the anagen-to-catagen/telogen (A:C/T) ratio. These parameters were assessed using phototrichoscopy and phototrichogram via TrichoScan®. The study was approved by an ethics committee and conducted by two independent board-certified dermatologists at two study sites.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40 years
* Sex: female
* Telogen effluvium diagnosis with hair loss > 100 hairs, confirmed using validated "modified wash test"
* Otherwise, healthy volunteers
* Refraining from systemic, topical, oral products with similar effects to the active product
* Signed informed consent
* Maintenance of daily cosmetic and dietary routine
* Availability to attend all visits
* Compliance with all protocol requirements

Exclusion Criteria:

* Previous use of active product
* Participation in similar studies or usage of anti-hair loss products within the last 3 months
* History of dermatological treatment (e.g. mesotherapy) and/or hair transplant
* Skin or scalp diseases (e.g. psoriasis, dermatitis, alopecias)
* Alopecia secondary to medical diseases (e.g. hypothyroidism, anemia)
* Ongoing treatment for or diagnosis of systemic disease
* Hormonal treatment (oral or topical contraceptives) within 6 months prior to study start
* Known allergy or intolerance, including to any of the ingredients of the active product
* Pregnancy, post-partum (6 months) or breastfeeding

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Increase in hair density | From enrollment to the end of treatment at 180 days.
  From phototrichogram on the temporoparietal area of the scalp.

SECONDARY OUTCOMES:
Change in the Anagen-to-Catagen/Telogen ratio | From enrollment to the end of treatment at 180 days.
  From phototrichogram on the temporoparietal area of the scalp.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Zurko-CTC, Barcelona
  - Clínica AB Derma, Madrid

REFERENCES:
- [Derived] Bernardez C, Podlipnik S, Westgate GE, Paus R, Zamfir L, Grohmann D, Saez Moya M. Efficacy and Safety of a Drinkable Nutraceutical in Premenopausal Women with Telogen Effluvium: A 6-Month, Randomized, Multicenter, Double-Blind, Placebo-Controlled Study. Dermatol Ther (Heidelb). 2025 Nov 25. doi: 10.1007/s13555-025-01585-x. Online ahead of print. PMID 41288927